CLINICAL TRIAL: NCT02011919
Title: Treatment of Breast Fibroadenoma With High Intensity Focused Ultrasound (HIFU)
Acronym: HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU / TU / FA
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echopulse (Other): Echopulse HIFU
  Interventions: Device: Echopulse

INTERVENTIONS:
Device: Echopulse — HIFU Under ultrasound guidance

SUMMARY:
This is a monocenter, open-label, uncontrolled study in accordance with §23b MPG to evaluate the efficacy of the HIFU-treatment of fibroadenoma using the TH-One device

Objectives Primary objective: To evaluate the efficacy of HIFU in the treatment of the breast fibroadenoma using the TH-One device Secondary objective: To evaluate the tolerability of the HIFU using the TH-One device

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older with at least one diagnosed breast fibroadenoma.
* Diagnosis of fibroadenoma must be based on:

  * clinical examination,
  * women ≤ 40 years of age: ultrasound image alone; women > 40 years of age: ultrasound image and mammogram,
  * histological confirmation of fibroadenoma of the breast.
* Patient's fibroadenoma size as determined by ultrasound imaging: the longest diameter is limited to 25 mm.
* Women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to HIFU treatment.
* Patient must be able to understand the nature and the extent of the study and the procédures required and be willing and able to complete the screening and study procedures.
* Patient must give written informed consent (personally signed and dated) before completing any study-related procedure.

Exclusion Criteria:

* Patient who is pregnant or breast-feeding.
* Patient with history of ipsilateral breast cancer within 5 years prior to study inclusion or radio therapy to the target breast within 5 years prior to study inclusion.
* Patient with implant on the treated breast.
* Patient with target fibroadenoma pre-treated by cryoablation or interstitial laser therapy within 12 month before recruiting for HIFU.
* Patient's fibroadenoma not clearly visible on the ultrasound images (in B mode) at the inclusion visit.
* Patient participating in other studies using drugs or medical devices within 3 months prior to study inclusion or during study participation including the follow-up period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
FA volume changes from baseline | Every year during 5 years

SECONDARY OUTCOMES:
Palpability | Every year during 5 years
  Lack of palpable lesion
Pain assessment | Every year during 5 years
  Pain free if pain at baseline (pain related to the FA)
Cosmetic result | Every year during 5 years
  Cosmetic result (as judged by investigator)
Gland vascularisation | Every year during 5 years
  Gland vascularisation (compared to baseline) power Doppler at day 7, month 6 and 12, year 2, 3, 4 and 5 after the HIFU session
Histological outcome | Every year during 5 years
  Histological outcome through core needle biopsy after 12 month
Energy settings | Every year during 5 years
  Energy setting to obtain reduction in volume or total regression of the FA at 12 months, 2, 3, 4 and 5 years follow-up
Breast immobilization | Every year during 5 years
  Quality and ease of use of breast immobilization
Duration of the treatment session | Every year during 5 years
  Duration of the treatment session (min)
Ease of implementation of treatment | Every year during 5 years
  Ease of implementation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tubingen University Hospital, Tübingen, Germany

REFERENCES:
- [Derived] Hahn M, Fugunt R, Schoenfisch B, Oberlechner E, Gruber IV, Hoopmann U, Roehm C, Helms G, Taran FA, Hartkopf AD, Warzecha H, Wiesinger B, Brucker SY, Boeer B. High intensity focused ultrasound (HIFU) for the treatment of symptomatic breast fibroadenoma. Int J Hyperthermia. 2018;35(1):463-470. doi: 10.1080/02656736.2018.1508757. Epub 2018 Sep 11. PMID 30204024